CLINICAL TRIAL: NCT04389879
Title: CAD/CAM Fixed Retainers vs. Conventional Multistranded Fixed Retainers in Orthodontic Patients. Comparison of Stability, Retainer Failure Rate, Adverse Effects, Cost-effectiveness, and Patient Satisfaction. A Randomized Controlled Clinical Trial.
Acronym: Retention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 01286
Record Dates: First submitted 2020-04-16; First posted 2020-05-15 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Relapse
Keywords: Orthodontic retainer; relapse; stability; CAD/CAM; fixed retainer
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Two-center randomized controlled clinical trial. Consecutive patients who are about to finish their fixed appliance orthodontic treatment at the two orthodontic departments will be screened for eligibility criteria. Eligible subjects will be randomized to have one of either two different fixed retainers to be bonded (to the upper and lower anterior teeth) by one operator in each center.
  Subjects will be allocated 1:1 into one of the two groups.
Masking Description: The outcome assessor will be blinded only to the patient satisfaction and cost-effectiveness outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM (Experimental): CAD/CAM custom-cut Nickel Titanium (NiTi) FR
  Interventions: Other: Bonding of either CAD/CAM or conventional multistranded stainless steel fixed retainer
- Conventional multistranded (Active Comparator): Conventional multistranded Stainless Steel (SS) FR
  Interventions: Other: Bonding of either CAD/CAM or conventional multistranded stainless steel fixed retainer

INTERVENTIONS:
Other: Bonding of either CAD/CAM or conventional multistranded stainless steel fixed retainer — Investigate and compare the clinical effectiveness of two types of fixed retainers; CAD/CAM vs. multistranded wire.

SUMMARY:
Introduction:

Orthodontic retainers are used after the completion of orthodontic treatment to assure dental occlusal stability and to maintain the achieved end-result. However, without retention teeth could go back to their initial dental malposition or could even take a different unpredicted position resulting once again in dental malocclusion (a deviation from normal occlusion).

There are different types of retainers, some are fixed (glued to the back of the front teeth), and others are removable (can be removed and replaced into the mouth by the patient).

While there are various retainers used for retention (stability), there is no perfect method. Fixed retainers (FRs) are used worldwide. On the one hand, FRs focus on preventing relapse. On the other hand, there are sometimes some adverse effects of retainers; they could fail at a certain point (break/get loose), or cause unwanted tooth movements. Until now, the choice of a retention method is based solely on clinicians' experience as there is no substantial evidence regarding the best retention method or the duration of the retention period. Some clinicians prolong the retention period while others prefer to keep the retainers for an indefinite time.

As the world is advancing, so is the orthodontic science. New FR fabricated by CAD/CAM (Computer-Aided Design/Computer-Aided Manufacturing), are assumed to have greater accuracy, better fit, and most importantly, might offer a passive positioning of the retainer. However, the evidence about CAD/CAM FRs is very limited.

Purpose:

To investigate and compare the clinical effectiveness of two types of FRs; CAD/CAM vs. multistranded wire, in terms of stability (primary outcome), failure rate, adverse effects, cost-effectiveness, and patient satisfaction (secondary outcomes), substantial up to 5 years after retainer placement.

Hypotheses:

Compared to traditional multistranded FRs, CAD/CAM FRs have:

* Better long term stability,
* Similar failure rate,
* Fewer adverse effects,
* Similar cost-effectiveness and patient satisfaction.

DETAILED DESCRIPTION:
Material and Methods

Setting: Section of Orthodontics, Department of Dentistry and Oral Health, Aarhus University, Denmark and Department of Orthodontics, Faculty of Dentistry, University of Oslo, Norway.

Sample size: 126 participants are needed for this study.

Randomization: After oral and written consent is obtained, allocation to groups, either conventional multistranded Stainless Steel fixed retainers, or CAD/CAM custom-cut Nickel Titanium fixed retainers, will take place at the last appointment before debonding. Subjects will be allocated 1:1 into one of the two groups.

Intervention protocol: After completing a full active orthodontic treatment, at both centers. The achieved treatment end result has to be maintained in the long term in order to prevent relapse (movement of teeth to the initial malocclusion). One of either two different fixed retainers will be bonded (to the upper and lower anterior teeth) by one operator in each center.

This study follows a standard retention protocol procedure carried at both centers and has a long term posttreatment follow-up of 5 years. Patients will be recalled for follow-up appointments after 1, 3, 6, 12, 24, 36 and 60 months. At follow-up visits, we will perform the following: at 1, and 3 months - a clinical examination. At 6, 12, 24, 36, and 60 months - a clinical examination, a digital impression of the teeth known as "an intraoral scan" (Trios 3, 3Shape, Copenhagen, Denmark) and intraoral photographs. In addition, at 1, 6, and 12 months patients will be asked to fill out a Visual Analogue Scale (VAS) form regarding patient satisfaction Furthermore, we will investigate stability by superimposition (Orthoanalyzer, 3Shape, Copenhagen, Denmark) together with recording of adverse effects (i.e. any changes in torque and/or rotations of the teeth).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients.
2. Age: 12-25 years old (at time of debonding).
3. Presence of all maxillary and mandibular anterior teeth, with normal shape and size.
4. Completion of a course of fixed appliance therapy involving both dental arches.
5. Subjects willing to consent to the trial and comply with the trial regime.

No restriction to presenting initial malocclusion, type of active orthodontic treatment undertaken provided that it included full fixed appliances (functional/removable appliances in combination with fixed appliances - extraction or non-extraction)

Exclusion Criteria:

1. Patients with cleft lip or palate, or both or any other craniofacial syndrome.
2. Patients who had surgical correction of the jaws: Le fort I (2- or 3-piece maxilla) or SARPE (surgically assisted rapid palatal expansion).
3. Lingual appliance treatments.
4. Periodontal disease.
5. Hypoplasia of enamel.
6. Fluorosis.
7. Active caries, restorations or fractures in the anterior teeth.
8. Patients who have had separate debonding appointments for each jaw, with a difference of more than 2 months in between.
9. Re-treated patients.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stability | From debonding (T1), and after 6, 12, 24, 36 and 60 months in retention phase (T4, T5, T6, T7, and T8 respectively)
  Change in lower incisor crowding will be assessed using Little's Irregularity Index (LII). Change in overall occlusal stability will be assessed by the Peer Assessment Rating (PAR) index. In addition, changes in arch dimensions, occlusal relationships, and re-opening of extraction spaces will be recorded.

SECONDARY OUTCOMES:
Failure rate and survival time | From the time of retainer bonding to the first failure episode: From debonding, and up to 60 months later
  Calculated from the first day of retainer's bonding to the day of the first failure episode
Adverse effects | From debonding, and up to 60 months later
  Screen for unexpected posttreatment changes in the mandibular anterior region associated with the use of both types of fixed retainers
Cost-effectiveness | From debonding, and up to 60 months later
  Unit costs in euros (€) will be used to value the resources included
Patient satisfaction | From debonding, and after 1, 6 and 12 months in retention phase
  Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Cornelis, Principal Investigator — University of Aarhus
Locations (2):
- Marie Anne Michele Cornelis, Aarhus, Denmark
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owman G, Bjerklin K, Kurol J. Mandibular incisor stability after orthodontic treatment in the upper arch. Eur J Orthod. 1989 Nov;11(4):341-50. doi: 10.1093/oxfordjournals.ejo.a036005. PMID 2591482
- [Background] Al Yami EA, Kuijpers-Jagtman AM, van 't Hof MA. Stability of orthodontic treatment outcome: follow-up until 10 years postretention. Am J Orthod Dentofacial Orthop. 1999 Mar;115(3):300-4. doi: 10.1016/s0889-5406(99)70333-1. PMID 10066979
- [Background] Littlewood SJ, Millett DT, Doubleday B, Bearn DR, Worthington HV. Retention procedures for stabilising tooth position after treatment with orthodontic braces. Cochrane Database Syst Rev. 2004;(1):CD002283. doi: 10.1002/14651858.CD002283.pub2. PMID 14973985
- [Background] Reitan K. Clinical and histologic observations on tooth movement during and after orthodontic treatment. Am J Orthod. 1967 Oct;53(10):721-45. doi: 10.1016/0002-9416(67)90118-2. No abstract available. PMID 5233926
- [Background] Little RM, Wallen TR, Riedel RA. Stability and relapse of mandibular anterior alignment-first premolar extraction cases treated by traditional edgewise orthodontics. Am J Orthod. 1981 Oct;80(4):349-65. doi: 10.1016/0002-9416(81)90171-8. PMID 6945805
- [Background] Littlewood SJ, Millett DT, Doubleday B, Bearn DR, Worthington HV. Orthodontic retention: a systematic review. J Orthod. 2006 Sep;33(3):205-12. doi: 10.1179/146531205225021624. PMID 16926314
- [Background] Gardner SD, Chaconas SJ. Posttreatment and postretention changes following orthodontic therapy. Angle Orthod. 1976 Apr;46(2):151-61. doi: 10.1043/0003-3219(1976)0462.0.CO;2. PMID 1064343
- [Background] Goldberg AI, Behrents RG, Oliver DR, Buschang PH. Facial divergence and mandibular crowding in treated subjects. Angle Orthod. 2013 May;83(3):381-8. doi: 10.2319/061912-505.1. Epub 2012 Oct 18. PMID 23075061
- [Background] Artun J, Spadafora AT, Shapiro PA. A 3-year follow-up study of various types of orthodontic canine-to-canine retainers. Eur J Orthod. 1997 Oct;19(5):501-9. doi: 10.1093/ejo/19.5.501. PMID 9386336
- [Background] Bolla E, Cozzani M, Doldo T, Fontana M. Failure evaluation after a 6-year retention period: a comparison between glass fiber-reinforced (GFR) and multistranded bonded retainers. Int Orthod. 2012 Mar;10(1):16-28. doi: 10.1016/j.ortho.2011.12.005. Epub 2012 Jan 11. English, French. PMID 22240271
- [Background] Rose E, Frucht S, Jonas IE. Clinical comparison of a multistranded wire and a direct-bonded polyethylene ribbon-reinforced resin composite used for lingual retention. Quintessence Int. 2002 Sep;33(8):579-83. PMID 12238688
- [Background] Salehi P, Zarif Najafi H, Roeinpeikar SM. Comparison of survival time between two types of orthodontic fixed retainer: a prospective randomized clinical trial. Prog Orthod. 2013 Sep 11;14:25. doi: 10.1186/2196-1042-14-25. PMID 24326013
- [Background] Saleh M, Hajeer MY, Muessig D. Acceptability comparison between Hawley retainers and vacuum-formed retainers in orthodontic adult patients: a single-centre, randomized controlled trial. Eur J Orthod. 2017 Aug 1;39(4):453-461. doi: 10.1093/ejo/cjx024. PMID 28430890
- [Background] Hichens L, Rowland H, Williams A, Hollinghurst S, Ewings P, Clark S, Ireland A, Sandy J. Cost-effectiveness and patient satisfaction: Hawley and vacuum-formed retainers. Eur J Orthod. 2007 Aug;29(4):372-8. doi: 10.1093/ejo/cjm039. PMID 17702797
- [Background] Tynelius GE, Lilja-Karlander E, Petren S. A cost-minimization analysis of an RCT of three retention methods. Eur J Orthod. 2014 Aug;36(4):436-41. doi: 10.1093/ejo/cjt070. Epub 2013 Oct 1. PMID 24084630
- [Background] Forde K, Storey M, Littlewood SJ, Scott P, Luther F, Kang J. Bonded versus vacuum-formed retainers: a randomized controlled trial. Part 1: stability, retainer survival, and patient satisfaction outcomes after 12 months. Eur J Orthod. 2018 Jul 27;40(4):387-398. doi: 10.1093/ejo/cjx058. PMID 29059289
- [Background] Wolf M, Schumacher P, Jager F, Wego J, Fritz U, Korbmacher-Steiner H, Jager A, Schauseil M. Novel lingual retainer created using CAD/CAM technology: evaluation of its positioning accuracy. J Orofac Orthop. 2015 Mar;76(2):164-74. doi: 10.1007/s00056-014-0279-8. English, German. PMID 25744094
- [Background] Jost-Brinkmann PG, Cacciafesta V, Miethke RR. Computer-aided fabrication of bonded lingual retainers. J Clin Orthod. 1996 Oct;30(10):559-63. No abstract available. PMID 10356474
- [Background] Artun J, Zachrisson B. Improving the handling properties of a composite resin for direct bonding. Am J Orthod. 1982 Apr;81(4):269-76. doi: 10.1016/0002-9416(82)90212-3. PMID 6217753
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332
- [Background] Bjering R, Sandvik L, Midtbo M, Vandevska-Radunovic V. Stability of anterior tooth alignment 10 years out of retention. J Orofac Orthop. 2017 Jul;78(4):275-283. doi: 10.1007/s00056-017-0084-2. Epub 2017 Apr 13. PMID 28409195
- [Background] Renkema AM, Renkema A, Bronkhorst E, Katsaros C. Long-term effectiveness of canine-to-canine bonded flexible spiral wire lingual retainers. Am J Orthod Dentofacial Orthop. 2011 May;139(5):614-21. doi: 10.1016/j.ajodo.2009.06.041. PMID 21536204
- [Background] Katsaros C, Livas C, Renkema AM. Unexpected complications of bonded mandibular lingual retainers. Am J Orthod Dentofacial Orthop. 2007 Dec;132(6):838-41. doi: 10.1016/j.ajodo.2007.07.011. PMID 18068606
- [Background] Pazera P, Fudalej P, Katsaros C. Severe complication of a bonded mandibular lingual retainer. Am J Orthod Dentofacial Orthop. 2012 Sep;142(3):406-9. doi: 10.1016/j.ajodo.2012.01.019. PMID 22920708
- [Derived] Pullisaar H, Cattaneo PM, Gera A, Sankiewicz M, Bilinska M, Vandevska-Radunovic V, Cornelis MA. Stability, survival, patient satisfaction, and cost-minimization of CAD/CAM versus conventional multistranded fixed retainers in orthodontic patients: a 2-year follow-up of a two-centre randomized controlled trial. Eur J Orthod. 2024 Apr 1;46(2):cjae006. doi: 10.1093/ejo/cjae006. PMID 38394353
- [Derived] Gera A, Pullisaar H, Cattaneo PM, Gera S, Vandevska-Radunovic V, Cornelis MA. Stability, survival, and patient satisfaction with CAD/CAM versus conventional multistranded fixed retainers in orthodontic patients: a 6-month follow-up of a two-centre randomized controlled clinical trial. Eur J Orthod. 2023 Feb 10;45(1):58-67. doi: 10.1093/ejo/cjac042. PMID 35964235